CLINICAL TRIAL: NCT06260410
Title: Data Collection in Lutetium Treated Prostate Cancer: Recording of Progression and Tumor Characteristics
Acronym: LUTRAC
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, S. L. W. (Stijn) Koolen, Assistant Professor, Hospital Pharmacist, Clinical Pharmacologist, Erasmus Medical Center
Other Study IDs: 10512; NL84672.078.23 (Other: CCMO)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer Metastatic
Keywords: mCRPC; Lu-PSMA; Prostate Cancer; Radioligand Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor DNA is obtained as part of this study to explore PSMA expression and how this relates to therapy outcomes. Plasma samples are stored according to standard of conservation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Blood draw for ctDNA and circulating tumor cell collection. — During routine blood sample collection, additional blood will be drawn for analysis of ctDNA and to collect Circulating Tumor Cells.

SUMMARY:
This prospective study aims to collect data and blood biomarkers from patients undergoing Lu-PSMA therapy at the Erasmus MC. In doing so, it will provide real-world efficacy and safety data on the drug, gather dosimetry data and explore putative biomarkers to identify patients who most benefit from Lu-PSMA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be at least 18 years old.
* Participants should be able to understand the written information and be able to provide informed consent.
* Participants are planned to start treatment with Lu-PSMA as a part of regular clinical care.

Exclusion Criteria:

None applicable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic castration resistant prostate cancer set to receive treatment with Lutetium-177 Prostate Specific Membrane Antigen (Lu-PSMA) as a part of regular clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 44 months
  Overall survival will be defined as the time from inclusion to death from any cause.

SECONDARY OUTCOMES:
Progression free survival | 44 months
  Progression free survival will be defined as clinical, radiological or PSA progression according to Prostate Cancer Working Group 3 (PCWG3) or death, whichever occurs first.
Heterogeneity of PSMA-positivity | 44 months
  Exploring heterogeneity of PSMA-positivity in circulating tumor cells (CTC) prior to treatment with Lutetium-PSMA.
Effect of CTC PSMA expression on response to treatment. | 44 months
  Exploring whether there is an association between the fraction of PSMA positive CTCs and response to Lutetium-PSMA treatment.
Effect of biomarkers in blood on response to treatment. | 44 months
  Exploring the association between biomarkers in blood and response to treatment
PSMA-PET scan data and response to treatment. | 44 months
  Exploring associations between PSMA-PET and therapy scans and response to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands